CLINICAL TRIAL: NCT02856594
Title: Minimizing ICU Neurological Dysfunction With Dexmedetomidine-induced Sleep (MINDDS): A Randomized Placebo-controlled Trial
Brief Title: Minimizing ICU Neurological Dysfunction With Dexmedetomidine-induced Sleep
Acronym: MINDDS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Oluwaseun Johnson-Akeju, MD, MMSc, Assistant Professor in Anesthesia, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016P000742; 1R01AG053582 (NIH)
Record Dates: First submitted 2016-07-29; First posted 2016-08-05 (Estimated); Results first posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-02

CONDITIONS: Postoperative Delirium; Sleep; Anesthesia
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine-induced sleep (Experimental): Precedex (Dexmedetomidine) intervention: Intravenous administration of 1mcg/kg over 40 minutes.
  Interventions: Drug: Dexmedetomidine
- Placebo (Placebo Comparator): Placebo of normal saline: Intravenous administration of normal saline over 40 minutes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine
  Other Names: Precedex
  Arms: Dexmedetomidine-induced sleep
Drug: Placebo — Placebo
  Other Names: Normal Saline
  Arms: Placebo

SUMMARY:
This study aims to determine whether, compared with placebo, the nighttime administration of a intravenous dexmedetomidine is effective at inducing sleep and preventing postoperative delirium in extubated post-cardiac surgical patients.

DETAILED DESCRIPTION:
Delirium is an acute brain dysfunction characterized by disturbances in attention, awareness, and cognition not explained by a preexisting neurocognitive disorder. Although the increased mortality rates ascribed to delirium remain debatable, delirium remains a leading cause of preventable morbidity in hospitalized elderly patients. It is also associated with prolonged hospitalization, prolonged institutionalization, and long-term cognitive deficits. Patients with pre-existing dementia, such as Alzheimer's disease, are especially vulnerable to developing delirium. The total healthcare cost attributable to delirium is estimated between $143 and $152 billion annually. In the United States, delirium occurs in approximately 80% of critically ill patients admitted to medical/surgical intensive care units (ICU), and 15% of patients admitted to cardiac surgical (CS) ICU. Most patients diagnosed with delirium also present with multiple comorbidities (sepsis, multi-organ failure) that significantly confound our understanding of this disease. Thus, to date, no pharmacological intervention to treat delirium has been identified.

There is mounting evidence to suggest that sleep deprivation may be a modifiable risk factor for the development of delirium. Presently, pharmacological treatment with no current medication (benzodiazepines, antipsychotics) induces natural sleep or reliably reduces the incidence of delirium. The investigators have found that biomimetic sleep, defined here as pharmacological induction of rapid eye movement sleep (REM) and non-REM (N1, N2, N3) sleep states using dexmedetomidine, can now be achieved in humans. The overall objective of this study is to evaluate the efficacy of biomimetic sleep in reducing the incidence and severity of delirium in extubated CSICU patients. The investigators will also assess for peri-operative electroencephalogram biomarkers of delirium, and the association between delirium and chronic neuroinflammation using positron emission tomography. The MINDDS study is poised to enable therapeutic and diagnostic discoveries to aid the care of elderly patients who are at risk for developing postoperative delirium.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60
* Scheduled for a cardiac surgical procedure with planned post-operative admission to the CSICU for ≥ 24 hours
* Scheduled same day surgical admission

Exclusion Criteria:

* Blind, deafness or the inability to speak English
* Greater than 2 days of ICU admission in the month preceding the current surgical procedure
* Renal and liver failure requiring dialysis or Child-Pugh score > 5
* Follow-up difficulties (i.e. active substance abuse, psychotic disorder, homelessness)
* Previous cardiac surgery within 1 year of surgical procedure
* Allergy to dexmedetomidine
* Chronic therapy with benzodiazepines and/or antipsychotics
* Severe deficit due to structural or anoxic brain damage
* Surgical procedure requiring total circulatory arrest

Objective Drop Criteria

* Scheduled for a second surgical procedure during hospital stay
* Post-operative intubation > 12 hours

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 469 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2022-02-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Immediately
Access Criteria: De-identified data and a data dictionary will be made available upon reasonable request to researchers who provide a methodologically sound proposal and whose use of the data has been approved the study authors. Data will be made available immediately following publication, with no anticipated end date, to achieve the aims specified in the approved proposal. Proposals should be directed to oluwaseun.akeju@mgh.harvard.edu.

REFERENCES:
- [Derived] Freedman IG, Boncompte G, Qu JZ, Khawaja ZQ, Turco I, Mueller A, Wiredu K, McKay TB, Westover MB, Pedemonte JC, Akeju O. Anesthesia-induced electroencephalogram oscillations and perioperative outcomes in older adults undergoing cardiac surgery. J Clin Anesth. 2025 Mar;102:111770. doi: 10.1016/j.jclinane.2025.111770. Epub 2025 Feb 7. PMID 39921932
- [Derived] Wiredu K, Mueller A, McKay TB, Behera A, Shaefi S, Akeju O. Sex Differences in the Incidence of Postoperative Delirium after Cardiac Surgery: A Pooled Analyses of Clinical Trials. Anesthesiology. 2023 Oct 1;139(4):540-542. doi: 10.1097/ALN.0000000000004656. No abstract available. PMID 37535937
- [Derived] Qu JZ, Mueller A, McKay TB, Westover MB, Shelton KT, Shaefi S, D'Alessandro DA, Berra L, Brown EN, Houle TT, Akeju O; MINDDS Study Team. Nighttime dexmedetomidine for delirium prevention in non-mechanically ventilated patients after cardiac surgery (MINDDS): A single-centre, parallel-arm, randomised, placebo-controlled superiority trial. EClinicalMedicine. 2022 Dec 24;56:101796. doi: 10.1016/j.eclinm.2022.101796. eCollection 2023 Feb. PMID 36590787
- [Derived] Shelton KT, Qu J, Bilotta F, Brown EN, Cudemus G, D'Alessandro DA, Deng H, DiBiasio A, Gitlin JA, Hahm EY, Hobbs LE, Houle TT, Ibala R, Loggia ML, Pavone KJ, Shaefi S, Tolis G, Westover MB, Akeju O. Minimizing ICU Neurological Dysfunction with Dexmedetomidine-induced Sleep (MINDDS): protocol for a randomised, double-blind, parallel-arm, placebo-controlled trial. BMJ Open. 2018 Apr 20;8(4):e020316. doi: 10.1136/bmjopen-2017-020316. PMID 29678977

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were no significant events in the study following enrollment but prior to assignment of participants to an arm or group. All enrolled subjects were assigned to either of the two study groups.
Period: Overall Study
Arm/Group | Dexmedetomidine-induced Sleep | Placebo
Started | 234 | 235
Analysis Population | 188 | 206
Completed | 188 | 206
Not Completed | 46 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine-induced Sleep | Placebo | Total
Number analyzed (Participants) | 188 | 206 | 394
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 59 | 49 | 108
  >=65 years | 129 | 157 | 286
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 67.5 [63.0 to 73.0] | 70.0 [65.0 to 75.0] | 69.0 [64.0 to 74.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 62 | 106
  Male | 144 | 144 | 288
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 179 | 194 | 373
  Unknown or Not Reported | 8 | 10 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 182 | 202 | 384
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Delirium Incidence at Baseline [Count of Participants; unit: Participants] | 0 | 0 | 0
Preoperative Cognitive Status [Median (Inter-Quartile Range); unit: score on a scale] — Telephone Montreal Cognitive Assessment
  score on a scale | 19.0 [17.0 to 20.0] | 19.0 [18.0 to 20.0] | 19.0 [17.0 to 20.0]
Preoperative Health Related Quality of Life [Median (Inter-Quartile Range); unit: Values are reported using a T-Score.] — PROMIS-29 questionnaires
  Values are reported using a T-Score.
    Global Health - Physical | 50.8 [42.3 to 57.7] | 50.8 [44.9 to 57.7] | 50.8 [42.3 to 57.7]
    Global Health - Mental | 56.0 [50.8 to 62.5] | 56.0 [48.3 to 62.5] | 56.0 [50.8 to 62.5]
    Physical Function | 44.6 [38.8 to 52.5] | 46.4 [40.1 to 52.5] | 45.5 [39.58 to 52.5]
    Pain Interference | 40.7 [40.7 to 55.4] | 40.7 [40.7 to 51.2] | 40.7 [40.7 to 53.2]
    Applied Cognition | 52.4 [45.9 to 62.7] | 51.2 [45.9 to 62.7] | 51.7 [45.9 to 62.7]
    Sleep Disturbance | 50.5 [43.8 to 56.1] | 50.5 [43.8 to 54.3] | 50.5 [43.8 to 56.1]

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Delirium
Description: Confusion Assessment Method
Time Frame: Post operative day 1 (24 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine-induced Sleep | Placebo
Number analyzed (Participants) | 175 | 189
Participants | 5 | 16
Statistical Analysis 1: Comparison: Dexmedetomidine-induced Sleep vs Placebo; Test type: Superiority; p = 0.029, Regression, Logistic; Odds Ratio (OR) = 0.32, 95% CI 2-sided [0.10 to 0.83]

2. Secondary Outcome: ICU Delirium/Coma-free Days
Description: Confusion Assessment Method
Time Frame: Up until postoperative day 3, or up until postoperative day 7 or discharge for patients who are delirious beyond postoperative day 5
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine-induced Sleep | Placebo
Number analyzed (Participants) | 160 | 177
Participants
  0 Days | 0 | 2
  1 Day | 6 | 7
  2 Days | 8 | 16
  3 Days | 146 | 152

3. Secondary Outcome: Severity of Delirium
Description: Confusion Assessment Method (CAM): Minimum Score=0, Maximum Score=19, Higher Scores: indicate increased severity of delirium
Time Frame: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Dexmedetomidine-induced Sleep | Placebo
Number analyzed (Participants) | 160 | 177
score on a scale | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 5.0]
Statistical Analysis 1: Comparison: Dexmedetomidine-induced Sleep vs Placebo; Test type: Superiority; p = 0.24, Regression, Linear; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.89 to 1.03]

4. Secondary Outcome: 30-day, 90-day, and 180-day Mortality
Description: 30-day, 90-day, and 180-day mortality
Time Frame: Up to postoperative day 180 (6 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine-induced Sleep | Placebo
Number analyzed (Participants) | 188 | 206
Participants
  In Hospital Mortality | 3 | 1
  30 Days | 3 | 1
  90 Days | 4 | 1
  180 Days | 4 | 4

5. Secondary Outcome: Postoperative Cognitive Status
Description: Telephone Montreal Cognitive Assessment (tMoCA): Minimum Score=0, Maximum Score=22, Higher Scores: indicate better cognitive function
Time Frame: 30 days, 90 days, and 180 days postoperatively
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Dexmedetomidine-induced Sleep | Placebo
Number analyzed (Participants) | 137 | 138
score on a scale
  30 Days | 20.0 [18.0 to 21.0] | 20.0 [19.0 to 21.0]
  90 Days | 20.0 [19.0 to 21.0] | 20.0 [19.0 to 21.0]
  180 Days | 20.0 [19.0 to 21.0] | 21.0 [19.0 to 22.0]

6. Secondary Outcome: Postoperative Health Related Quality of Life
Description: This included the PROMIS Global Health SF V.1.1, PROMIS Physical Function SF 8b V.1.2, PROMIS Pain Interference SF 8a V.1.0, PROMIS Applied Cognition Abilities SF 8a V.1.0, and PROMIS Sleep Disturbance SF 4A V.1.0, respectively. Scores from each assessment were converted to a T-score for analysis with a mean of 50 and a standard deviation of 10, with lower scores on the PROMIS Pain Interference SF and PROMIS Sleep Disturbance SF considered better, whereas higher scores on all other assessments were considered better.
Time Frame: 30 days, 90 days, and 180 days postoperatively
Measure: Median (Inter-Quartile Range); unit: T-Score
Arm/Group | Dexmedetomidine-induced Sleep | Placebo
Number analyzed (Participants) | 137 | 138
T-Score
  PROMIS Global Health - Physical (30 Days) | 50.8 [44.9 to 54.1] | 47.7 [42.3 to 54.1]
  PROMIS Global Health - Physical (90 Days) | 54.1 [47.7 to 59.8] | 54.1 [47.7 to 57.7]
  PROMIS Global Health - Physical (180Days) | 57.7 [50.8 to 61.9] | 54.1 [50.8 to 61.9]
  PROMIS Global Health - Mental (30 Days) | 59.0 [50.8 to 67.6] | 56.0 [50.8 to 62.5]
  PROMIS Global Health - Mental (90 Days) | 59.0 [53.3 to 67.6] | 62.5 [56.0 to 67.6]
  PROMIS Global Health - Mental (180 Days) | 62.5 [53.3 to 67.6] | 62.5 [53.3 to 67.6]
  PROMIS Physical Function (30 Days) | 49.9 [40.7 to 55.8] | 52.3 [40.7 to 58.1]
  PROMIS Physical Function (90 Days) | 40.7 [40.7 to 51.2] | 40.7 [40.7 to 49.9]
  PROMIS Physical Function (180 Days) | 40.7 [40.7 to 47.9] | 40.7 [40.7 to 40.7]
  PROMIS Pain Interference (30 Days) | 49.9 [40.7 to 55.8] | 52.3 [40.7 to 58.1]
  PROMIS Pain Interference (90 Days) | 40.7 [40.7 to 51.2] | 40.7 [40.7 to 49.9]
  PROMIS Pain Interference (180 Days) | 40.7 [40.7 to 47.9] | 40.7 [40.7 to 40.7]
  PROMIS Applied Cognition (30 Days) | 54.6 [48.6 to 62.7] | 53.0 [47.7 to 62.7]
  PROMIS Applied Cognition (90 Days) | 53.0 [49.5 to 62.7] | 54.6 [47.7 to 62.7]
  PROMIS Applied Cognition (180 Days) | 54.6 [47.7 to 62.7] | 54.6 [48.6 to 62.7]
  PROMIS Sleep Disturbance (30 Days) | 50.5 [43.8 to 56.1] | 50.5 [43.8 to 56.1]
  PROMIS Sleep Disturbance (90 Days) | 48.4 [43.8 to 52.4] | 48.4 [41.1 to 52.4]
  PROMIS Sleep Disturbance (180 Days) | 46.2 [41.1 to 51.5] | 46.2 [41.1 to 50.5]

7. Secondary Outcome: Blood Delirium Biomarkers
Description: Blood samples will be taken including whole blood, serum, TruCulture, and PAXgene to assess proteins, DNA, and RNA.
Time Frame: perioperative
Reporting Status: Not Posted

8. Secondary Outcome: EEG Delirium Biomarkers
Description: EEG burst suppression and alpha power will be analyzed for association with delirium.
Time Frame: intraoperative
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Length of Hospital Stay
Description: Medical Record Review
Time Frame: from postoperative day 0 until date of hospital discharge (no prespecified length possible)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Dexmedetomidine-induced Sleep | Placebo
Number analyzed (Participants) | 188 | 206
days | 6.0 [5.0 to 8.0] | 6.0 [5.0 to 7.0]

ADVERSE EVENTS:
Time Frame: Adverse events were evaluated until discharge from the hospital. Mortality was assessed until 180 days postoperatively.
Description: Adverse events were collected via review of the electronic medical record or by phone call at 30, 90 or 180 days.
Arm/Group | Dexmedetomidine-induced Sleep | Placebo
All-Cause Mortality (participants affected / at risk) | 4/188 | 4/206
Serious Adverse Events (participants affected / at risk) | 0/188 | 0/206
Other Adverse Events (participants affected / at risk) | 0/188 | 0/206

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT02856594/Prot_SAP_000.pdf